CLINICAL TRIAL: NCT05781620
Title: Effects of Vitamin D Supplementation on Biochemical Reaction and Skeletal Muscle Synthesis in Prolonged Endurance Exercise and Cluster Set Configurations of Resistance Training
Brief Title: Vitamin D Supplementation in Healthy Adults in Prolonged Endurance Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: Panion & BF Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202205045; NSTC111-2410-H-038 -015 (Other Grant/Funding Number: National Science and Technology Council)
Record Dates: First submitted 2023-02-20; First posted 2023-03-23 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: An independent samples and dose titration design will be used to assign participants to the experimental group or placebo group.
Who Masked: Participant, Investigator
Masking Description: A double-blind, matched-pair study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental)
  Interventions: Dietary Supplement: Vitamin D
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Medium-chain triglycerides

INTERVENTIONS:
Dietary Supplement: Vitamin D — Participants received 5,000 IU of vitamin D orally twice daily for 4 weeks. If the serum 25(OH)D concentration exceeds 48 ng/mL, the intervention remains the same. However, if the serum 25(OH)D concentration is under 48 ng/mL, the dosage would increase by 2,500 IU. The principle remains the same at week 6.
  Arms: Vitamin D group
Dietary Supplement: Medium-chain triglycerides — Participants received the same amount of placebo matching vitamin D orally twice daily.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to investigate the effects of vitamin D supplementation on biochemistry response and skeletal muscle synthesis in prolonged endurance exercise.

DETAILED DESCRIPTION:
Endurance exercise mode will be used to evaluate the effects of vitamin D supplementation on cardiac biomarkers, metabolic hormones, oxidative damage, and inflammation responses. An independent samples and dose titration design will be used to assign 30 participants to the experimental group (n = 15) or placebo group (n = 15). All participants in the experimental group will have serum 25(OH)D concentrations higher than 48 ng/mL after supplementation period. After the prolonged endurance exercise test, the blood samples will be collected for analyzing biomarkers. Data will be analyzed by Two-way mixed design ANOVA.

ELIGIBILITY:
Inclusion criteria:

* The volunteers included have conditions as stated below :

  1. male adult between 20-40 years old without any history of cardiovascular, liver, kidney and diabetes disease
  2. no acute sport injury
  3. male adult whose concentration of 25(OH)D is under 30 ng/mL, and maximal oxygen consumption is over 40 ml/kg/min
  4. did not participated in any clinical trials or research in the last 3 months before our experiment
  5. no supplements were taken during the experimental period
  6. were requested to maintain their regular daily life style and avoid alcohol intake

Exclusion Criteria:

* The volunteers were excluded if they have the situation stated below:

  1. history of cardiovascular, liver, kidney and diabetes disease
  2. acute sport injury
  3. their concentration of 25(OH)D is over 30 ng/mL, or maximal oxygen consumption is under 40 ml/kg/mint
  4. participated in any clinical trials or experimental research in the last 3 months before our experiment
  5. taking supplement during the experimental period
  6. did not maintain their regular eating habit or drink alcohol

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Concentration of NT-proBNP | before exercise
Concentration of NT-proBNP | immediately after exercise
Concentration of NT-proBNP | 2-hour after exercise
Concentration of NT-proBNP | 24-hour after exercise
Concentration of cTnI | before exercise
Concentration of cTnI | immediately after exercise
Concentration of cTnI | 2-hour after exercise
Concentration of cTnI | 24-hour after exercise
Concentration of CK-MB | before exercise
Concentration of CK-MB | immediately after exercise
Concentration of CK-MB | 2-hour after exercise
Concentration of CK-MB | 24-hour after exercise
Concentration of CK | before exercise
Concentration of CK | immediately after exercise
Concentration of CK | 2-hour after exercise
Concentration of CK | 24-hour after exercise
Concentration of Testosterone | before exercise
Concentration of Testosterone | immediately after exercise
Concentration of Testosterone | 2-hour after exercise
Concentration of Testosterone | 24-hour after exercise
Concentration of Cortisol | before exercise
Concentration of Cortisol | immediately after exercise
Concentration of Cortisol | 2-hour after exercise
Concentration of Cortisol | 24-hour after exercise
Concentration of β-endorphin | before exercise
Concentration of β-endorphin | immediately after exercise
Concentration of β-endorphin | 2-hour after exercise
Concentration of β-endorphin | 24-hour after exercise
Concentration of Growth hormone | before exercise
Concentration of Growth hormone | immediately after exercise
Concentration of Growth hormone | 2-hour after exercise
Concentration of Growth hormone | 24-hour after exercise
Concentration of IGF-1 | before exercise
Concentration of IGF-1 | immediately after exercise
Concentration of IGF-1 | 2-hour after exercise
Concentration of IGF-1 | 24-hour after exercise
Concentration of TBARS | before exercise
Concentration of TBARS | immediately after exercise
Concentration of TBARS | 2-hour after exercise
Concentration of TBARS | 24-hour after exercise
Concentration of PC | before exercise
Concentration of PC | immediately after exercise
Concentration of PC | 2-hour after exercise
Concentration of PC | 24-hour after exercise
Concentration of SOD | before exercise
Concentration of SOD | immediately after exercise
Concentration of SOD | 2-hour after exercise
Concentration of SOD | 24-hour after exercise
Concentration of Catalase | before exercise
Concentration of Catalase | immediately after exercise
Concentration of Catalase | 2-hour after exercise
Concentration of Catalase | 24-hour after exercise
Concentration of TNF-α | before exercise
Concentration of TNF-α | immediately after exercise
Concentration of TNF-α | 2-hour after exercise
Concentration of TNF-α | 24-hour after exercise
Concentration of IL-8 | before exercise
Concentration of IL-8 | immediately after exercise
Concentration of IL-8 | 2-hour after exercise
Concentration of IL-8 | 24-hour after exercise
Concentration of IL-10 | before exercise
Concentration of IL-10 | immediately after exercise
Concentration of IL-10 | 2-hour after exercise
Concentration of IL-10 | 24-hour after exercise
Concentration of LDH | before exercise
Concentration of LDH | immediately after exercise
Concentration of LDH | 2-hour after exercise
Concentration of LDH | 24-hour after exercise
Concentration of IL-6 | before exercise
Concentration of IL-6 | immediately after exercise
Concentration of IL-6 | 2-hour after exercise
Concentration of IL-6 | 24-hour after exercise
Concentration of IL-15 | before exercise
Concentration of IL-15 | immediately after exercise
Concentration of IL-15 | 2-hour after exercise
Concentration of IL-15 | 24-hour after exercise
Concentration of leukocyte | before exercise
Concentration of leukocyte | immediately after exercise
Concentration of leukocyte | 2-hour after exercise
Concentration of leukocyte | 24-hour after exercise
Concentration of neutrophil | before exercise
Concentration of neutrophil | immediately after exercise
Concentration of neutrophil | 2-hour after exercise
Concentration of neutrophil | 24-hour after exercise
Concentration of eosinophil | before exercise
Concentration of eosinophil | immediately after exercise
Concentration of eosinophil | 2-hour after exercise
Concentration of eosinophil | 24-hour after exercise
Concentration of basophil | before exercise
Concentration of basophil | immediately after exercise
Concentration of basophil | 2-hour after exercise
Concentration of basophil | 24-hour after exercise
Concentration of monocyte | before exercise
Concentration of monocyte | immediately after exercise
Concentration of monocyte | 2-hour after exercise
Concentration of monocyte | 24-hour after exercise
Concentration of lymphocyte | before exercise
Concentration of lymphocyte | immediately after exercise
Concentration of lymphocyte | 2-hour after exercise
Concentration of lymphocyte | 24-hour after exercise
Concentration of CD4+ | before exercise
Concentration of CD4+ | immediately after exercise
Concentration of CD4+ | 2-hour after exercise
Concentration of CD4+ | 24-hour after exercise
Concentration of CD8+ | before exercise
Concentration of CD8+ | immediately after exercise
Concentration of CD8+ | 2-hour after exercise
Concentration of CD8+ | 24-hour after exercise
Concentration of CD19+ | before exercise
Concentration of CD19+ | immediately after exercise
Concentration of CD19+ | 2-hour after exercise
Concentration of CD19+ | 24-hour after exercise
Concentration of CD56+ | before exercise
Concentration of CD56+ | immediately after exercise
Concentration of CD56+ | 2-hour after exercise
Concentration of CD56+ | 24-hour after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan